CLINICAL TRIAL: NCT03919240
Title: CD19-targeting Chimeric Antigen Receptor T-cell Therapy for Patients with Refractory and Relapsed B-cell Acute Lymphoblastic Leukemia
Brief Title: CAR-T Cell Therapy Targeting to CD19 for R/R ALL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry); The Second People's Hospital of Huai'an (Other); Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ4601
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Acute Lymphoblastic Leukemia with Failed Remission
Keywords: Acute Lymphoblastic Leukemia; Refractory and relapsed; Chimeric antigen receptor T-cell therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR T-cell therapy (Experimental): Patients enrolled will receive infusion of CD19-targeting CART-cells
  Interventions: Biological: CAR T-cell therapy

INTERVENTIONS:
Biological: CAR T-cell therapy — Patients enrolled will receive infusion of CD19-targeting CAR T-cells with a target dose of 5~10×10E6/kg of recipient weight, after the preparative regimen consisted of fludarabin (30mg/m2, day -5 to -3) and cyclophosphamide (300mg/m2, day -5 to -3).

SUMMARY:
Refractory and relapsed (R/R) acute lymphoblastic leukemia (ALL) patients with active disease always have a dismal outcome. Chimeric antigen receptor (CAR) T-cell therapy targeting to Cluster of Differentiation Antigen 19 (CD19) has been proved as a potent approach to attain remission in B-cell R/R patients. Therefore, the investigators conduct atrial to evaluate the the efficacy and safety of locally producing CAR T cells targeting CD19, and to analyze the outcome of enrolled B-cell ALL patients with active disease or persistent residual disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as CD19+ B-cell acute lymphoblastic leukemia;
* Fail to achieve remission, or with persistent residual disease after at least 2 cycles of consolidation;
* With an estimated survival of higher than 3 months (according to investigator's judgement);
* Sufficient organ function: left ventricular ejection fractions≥ 0.5 by echocardiography, creatinine < 1.6 mg/dL, aspartate aminotransferase/aspartateaminotransferase < 3 x upper limit of normal, bilirubin <2.0 mg/dL;
* Karnofsky performance status ≥ 60 or ECOG ≤ 2.

Exclusion Criteria:

* Intolerant to immunosuppressive chemotherapies;
* With active infection or other uncontrolled complications;
* With history of seizure;
* Active hepatitis B or hepatitis C infection and HIV infection;
* Pregnant or lactating women, or patients refusing to take effective contraception measures;
* Other contraindications that considered inappropriate to participate in this trial (according to investigator's judgement).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Completeremission | 1 month post infusion
  defined as less than 5% blasts in the bone marrow without myelosuppression, no circulating blasts in peripheral blood, and the absence of extramedullary disease, regardless of cell count recovery
Minimal residual disease response | 1 month post infusion
  defined as less than 0.01% bone marrow blasts assessed by multiparameter flow cytometry, and absence of genetic aberrants assessed by karyotype analysis or molecular detection
Leukemia-free survival | 3 year post infusion
  calculating from the day of CAR T-cell infusion to death, disease progression or the end of follow-up

SECONDARY OUTCOMES:
Overall survival | 3 year post infusion
  calculating from the day of CAR T-cell infusion to death or the end of follow-up
Cumulative incidence of relapse | 3 year post infusion
  calculating from the day of CAR T-cell infusion to disease progression or the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The Fisrt Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Background] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Derived] Liu S, Zhang X, Dai H, Cui W, Yin J, Li Z, Yang X, Yang C, Xue S, Qiu H, Miao M, Chen S, Jin Z, Fu C, Li C, Sun A, Han Y, Wang Y, Yu L, Wu D, Cui Q, Tang X. Which one is better for refractory/relapsed acute B-cell lymphoblastic leukemia: Single-target (CD19) or dual-target (tandem or sequential CD19/CD22) CAR T-cell therapy? Blood Cancer J. 2023 Apr 24;13(1):60. doi: 10.1038/s41408-023-00819-5. PMID 37095120
- [Derived] Li M, Xue SL, Tang X, Xu J, Chen S, Han Y, Qiu H, Miao M, Xu N, Tan J, Kang L, Yu Z, Lou X, Xu Y, Chen J, Yan Z, Feng W, Wu D, Yu L. The differential effects of tumor burdens on predicting the net benefits of ssCART-19 cell treatment on r/r B-ALL patients. Sci Rep. 2022 Jan 10;12(1):378. doi: 10.1038/s41598-021-04296-3. PMID 35013456
- [Derived] Liu ZF, Chen LY, Wang J, Kang LQ, Tang H, Zhou Y, Zhou HX, Sun AN, Wu DP, Xue SL. Successful treatment of acute B lymphoblastic leukemia relapse in the skin and testicle by anti-CD19 CAR-T with IL-6 knocking down: a case report. Biomark Res. 2020 May 6;8:12. doi: 10.1186/s40364-020-00193-5. eCollection 2020. PMID 32399214